CLINICAL TRIAL: NCT05750303
Title: Circulating Serum VEGF, IGF-1 and MMP-9 and Expression of Their Genes as Potential Prognostic Markers of Recovery in Post-stroke Rehabilitation - Prospective Observational Study
Brief Title: Potential Prognostic Markers of Recovery in Post-stroke Rehabilitation
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Collaborators: University of Lodz (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNN/105/21/KE
Record Dates: First submitted 2023-02-02; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Ischemic Stroke
Keywords: stroke; recovery; biomarker; rehabilitation; VEGF; IGF-1; MMP-9
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subacute ischemic stroke: blood sample collection to determine VEGF, IGF-1 and MMP-9 level in plasma and expression of genes VEGF, IGF-1, MMP-9 in whole blood samples
- No ischemic stroke and no other neurological disease control group: blood sample collection to determine VEGF, IGF-1 and MMP-9 level in plasma and expression of genes VEGF, IGF-1, MMP-9 in whole blood samples

SUMMARY:
Despite increasingly effective early treatment strategies for ischemic stroke, post-stroke recovery is often incomplete and depend on spontaneous and therapeutic-induced processes related to neuroplasticity, angiogenesis and reperfusion. These processes are regulated by growth factors, neurotrophines, neurotransmitters, hormones and other factors. This study aims to search biomarkers that prognose brain repair ability and consequently estimate an outcome of stroke patients. The prognostic value of proteins VEGF, IGF-1 and MMP-9 and expression of genes VEGF, IGF-1, MMP-9 is evaluated in association with clinical scales including cognitive assessment scales and depression scales. Blood sample collection as well as scales recording are taken at baseline and 3 weeks later after rehabilitation.

DETAILED DESCRIPTION:
Despite increasingly effective early treatment strategies for ischemic stroke, post-stroke recovery is often incomplete and depend on spontaneous and therapeutic-induced processes related to neuroplasticity, angiogenesis and reperfusion. These processes are regulated by growth factors, neurotrophines, neurotransmitters, hormones and other factors. Recovery activity can be reflected both in the clinical assessment of the patient (based on the NIHSS or MRS scale for example) as well as on the biochemical and molecular level. This study aims to search biomarkers that prognose brain repair ability and consequently estimate an outcome of stroke patients. The prognostic value of proteins VEGF, IGF-1 and MMP-9 and expression of genes VEGF, IGF-1, MMP-9 is evaluated in association with clinical scales including cognitive assessment scales and depression scales. Furthermore, the collected data will be analyzed in relation to demographics and vascular risk factors. Blood sample collection as well as scales recording are taken at baseline and 3 weeks later after rehabilitation. The study group patients will undergo standard post-stroke rehabilitation programme provided by physiotherapist, every day for a period of 3 weeks with weekend gaps.

ELIGIBILITY:
Inclusion Criteria:

* subacute ischeamic stroke,
* age over 18,
* informed consent obtained

Exclusion Criteria:

* intracerebral haemorrhage,
* chronic or significant acute inflammatory factors,
* neurological illness other than ischeamic stroke,
* severe cardio-vascular disease like myocardial infarction less than 30 days, unstable angina pectoris,
* decompensated metabolic or endocrine diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subacute ischemic stroke patients received standard therapy
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
changes from baseline in IGF-1 level in plasma at 3 week of rehabilitation | baseline and 3 weeks later
  IGF-1 is a protein involved in neuroplasticity and angiogenesis processes. IGF-1 level in plasma - unit measure: ng/mL.
changes from baseline IGF-1 expression in whole blood sample at 3 week of rehabilitation | baseline and 3 weeks later
  IGF-1 is a protein involved in neuroplasticity and angiogenesis processes. IGF-1 mRNA gene expression is presented as -ΔCt
changes from baseline in VEGF level in plasma at 3 week of rehabilitation | baseline and 3 weeks later
  VEGF is a protein involved in neuroplasticity and angiogenesis processes. VEGF level in plasma - unit measure: pg/mL.
changes from baseline in VEGF expression in whole blood sample at 3 week of rehabilitation | baseline and 3 weeks later
  VEGF is a protein involved in neuroplasticity and angiogenesis processes. VEGF mRNA gene expression is presented as -ΔCt
changes from baseline in MMP-9 level in plasma at 3 week of rehabilitation | baseline and 3 weeks later
  MMP-9 is a protein involved in neuroplasticity and angiogenesis processes. MMP-9 level in plasma - unit of measure: pg/mL.
changes from baseline in MMP-9 expression in whole blood sample at 3 week of rehabilitation | baseline and 3 weeks later
  MMP-9 is a protein involved in neuroplasticity and angiogenesis processes. MMP-9 mRNA gene expression is presented as -ΔCt
changes form baseline in Mini Mental State Examination (MMSE) scale at 3-week rehabilitation | baseline and 3 weeks later
  Mini Mental State Examination is effective, screening tool for cognitive impairment, the maximum score for the MMSE is 30, a cut-off score of 23/24 (or below) indicates dementia, a score of 25 or higher is classed as normal
changes form baseline in The Geriatric Depression Scale (GDS) at 3-week rehabilitation | baseline and 3 weeks later
  The Geriatric Depression Scale is self-reported validated measure of depression in older adults, consists of 15 questions, users respond in a "Yes/No" format, scores 0-4 are considered normal, more than 5 indicate depression: 5-8 mild, 9-11 moderate and 12-15 severe depressive symptoms
changes form baseline in Barthel index scale at 3-week rehabilitation | baseline and 3 weeks later
  Barthel index is a scale used to measure performance in activities of daily living, the 10 items including the Barthel Index pay attention to self-care and mobility. Total possible scores range from 0 - 20, with lower scores indicating increased disability, a score of 17 represents normal ability.
changes form baseline in National Institutes of Health Stroke Scale (NIHSS) scale at 3-week rehabilitation | baseline and 3 weeks later
  National Institutes of Health Stroke Scale is a tool used to objectively quantify the impairment caused by stroke,total score ranging from 0 to 42 and the higher the score, the more severe the stroke
changes form baseline in Modified Rankin Scale (MRS) at 3-week rehabilitation | baseline and 3 weeks later
  Modified Rankin Scale measures degree of disability after stroke, ranges from grade 0 indicating a lack of symptoms to grade 6 indicating dead

CONTACTS AND LOCATIONS:
Overall Officials: Elzbieta Miller, Prof, Principal Investigator — Medical University of Lodz
Locations (1):
- Medical University of Lodz, Lodz, Poland